CLINICAL TRIAL: NCT05817383
Title: Blueberries, Gut Microbiota, and Metabolites in Depressed Older Adults - A Pilot Study
Brief Title: Berries, Bugs, and the Blues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Courtney Millar, Assistant Scientist I, Hebrew SeniorLife
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Pro00068528
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Depressive Symptoms
Keywords: Anthocyanins; Fiber; Aging
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freeze-dried Blueberry Powder (Experimental): Randomized participants will be asked to consume 48 grams of freeze-dried blueberry powder each day for 12 weeks.
  Interventions: Other: Freeze-dried Blueberry Powder
- Placebo Powder (Placebo Comparator): Randomized participants will be asked to consume 48 grams of a nutritionally matched placebo powder devoid of fiber and anthocyanins each day for 12 weeks.
  Interventions: Other: Placebo Powder

INTERVENTIONS:
Other: Freeze-dried Blueberry Powder — Participants will be asked to consume 48 grams of freeze-dried blueberry powder (~ equivalent to 2 cups of fresh blueberries) daily for 12 weeks. Participants will be asked to save any powder packet wrappers as a means to measure compliance. They will also be instructed to avoid consumption of foods/beverages that are high in anthocyanins and/or fiber.
  Arms: Freeze-dried Blueberry Powder
Other: Placebo Powder — Participants will be asked to consume 48 grams of a nutritionally matched placebo powder (that does not contain fiber or anthocyanins) daily for 12 weeks. Participants will be asked to save any powder packet wrappers as a means to measure compliance. They will also be instructed to avoid consumption of foods/beverages that are high in anthocyanins and/or fiber.
  Arms: Placebo Powder

SUMMARY:
This study aims to investigate the impact of daily freeze-dried blueberry powder consumption on the gut microbiota, fecal short chain fatty acids, and depressive symptom severity in 40older, sedentary adults with depressive symptoms.

DETAILED DESCRIPTION:
This study is an ancillary project to a currently funded randomized, placebo-controlled 12-week intervention in older, sedentary adults with depressive symptoms (IRB# Pro00064749). This specific project proposes distinct aims to the trial by gathering preliminary data on the synergistic impact of dietary fiber and anthocyanins (via freeze-dried blueberry powder) on the gut-microbiota, gut-derived metabolites, and depressive symptoms in older adults.

Participants will then be randomized to consume either 48 g of freeze-dried blueberry powder (~600 mg of anthocyanins and ~8 g of fiber) or 48 g of a nutritionally matched placebo powder (devoid of anthocyanins and fiber) each day for a total of 12 weeks.

At baseline, participants will be undergo assessments for depressive symptom severity and provide a fecal sample for gut microbiota and short chain fatty acid measurement. After 4, 8, and 12 weeks of consuming the powder there will be study visits that assess depressive symptom severity. Additionally, a final fecal sample will be taken after 12 weeks of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥65 years
* Self-reporting ≥ 8 hours of sitting per/day (e.g., sedentary behavior)
* Depressive symptoms (defined as ≥4 and <16 points on the center for epidemiological studies depression-scale

Exclusion Criteria:

* Unwilling to follow the study protocol
* A median daily step count >7,500 steps per day (as measured by the ActiGraph), or per discretion of the PI
* Cognitive impairment (defined as Montreal Cognitive Assessment, MoCA <22 points)
* Self-reporting a history of inflammatory bowel disease/syndrome, major depression, bipolar, schizophrenia, or other psychotic disorders, or per discretion of the PI
* Self-reporting type 1 or type 2 diabetes
* Allergic to intervention or control products
* Recent use (within the last 3 months) of antibiotics, or per discretion of the PI
* Recent use (within the last 3 months) of pro-biotics, or per discretion of the PI
* Current substance use disorder (Drug Abuse Screening Test, DAST-10>2 points)
* Current alcohol use disorder (Alcohol Use Disorders Identification Test - Consumption, AUDIT-C≥4 points)
* Unstable anti-depressant use (e.g., change in medication within last 3-6 months), or per discretion of the PI
* Current homicidal or suicidal ideation (assessed via the P4 Suicidality Screener)
* Current psychosis (via the Psychosis and Hallucinations Questionnaire, PHQ>12 points)
* Manic symptoms (assessed by the Mood Disorder Questionnaire, MDQ >5 points)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Millar, PhD, Principal Investigator — Hebrew SeniorLife, Marcus Institute of Aging, Harvard Medical Schools
Locations (1):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a sub-study of a larger, parent study (NCT 05735587) that aimed to recruit 40 individuals. All individuals that enrolled in the parent study (n=29) were offered to enroll in this sub study. Of the 29 individuals that enrolled in the parent study, 20 were enrolled in the sub-study. Of the 20 enrolled, 18 completed the sub-study.
Period: Overall Study
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (4) | 74 (6) | 73 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptom Severity
Description: Severity of depressive symptoms will be measured before and after the intervention with the Center for Epidemiological Studies Depression Scale-Revised (CESD-R). Scores range from 0 to 60 points, with higher scores indicating more sever depressive symptoms.
Time Frame: Change between baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder
Number analyzed (Participants) | 10 | 8
scores on a scale | -5 (3) | -4 (4)

2. Secondary Outcome: Abundance Microbes
Description: The abundance of the top 20 most prevalent microbes in our that produce short chain fatty acids (e.g., Bifidobacteria, Eubacterium, and Clostridium) will be evaluated by whole genome sequencing
Time Frame: Change between baseline and 12 week follow-up
Measure: Mean (Standard Deviation); unit: % Relative Abundance
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder
Number analyzed (Participants) | 10 | 8
% Relative Abundance | 1.28 (6.29) | 1.63 (11.65)

3. Secondary Outcome: Fecal Short Chain Fatty Acids (i.e., Butyrate)
Description: The relative abundance of short chain fatty acids (i.e., butyrate ) in feces will be measured using liquid chromatography mass spectrometry.
Time Frame: Percent change between baseline and 12 week follow-up
Measure: Mean (Standard Deviation); unit: Percent change of relative abundance
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder
Number analyzed (Participants) | 9 | 8
Percent change of relative abundance | -2 (48) | 27 (60)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the entire study intervention period for each participant which was approximately 12 weeks.
Arm/Group | Freeze-dried Blueberry Powder | Placebo Powder
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT05817383/Prot_SAP_001.pdf